CLINICAL TRIAL: NCT05825027
Title: A Risk Stratification Model for Health and Academic Outcomes in Children With Concussion Based on Novel Symptom Trajectory Typologies
Brief Title: Risk Stratification in Children With Concussion
Acronym: RSiCC
Status: Recruiting | Type: Observational
Sponsor: Duke University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Other Study IDs: Pro00111606; R01NS129617 (NIH)
Record Dates: First submitted 2023-04-10; First posted 2023-04-24 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Concussion, Brain; Mild Traumatic Brain Injury
MeSH Terms: conditions — Brain Concussion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This project will measure concussion symptoms, biological markers, and academic and social factors across the first year postconcussion to develop a model that enables early identification of and symptom management for children at higher risk for persistent postconcussive symptoms. Findings will provide novel insights into the longer-term effects of concussion on children's physical, psychological, and social well-being and support the development of personalized healthcare and school-based plans to reduce disparities in children's ability to return-to-learn and -play and improve postconcussion quality of life.

DETAILED DESCRIPTION:
Concussions occur at an alarming rate among U.S. schoolchildren, with one in five children experiencing a concussion by age 16. The number of children visiting emergency departments for concussions annually has increased by 50% over the past decade, with an estimated cost to the healthcare system of $1 billion/year. Compared to adults, children experience longer and more severe postconcussive symptoms (PCS). Severity and duration of PCS, however, vary considerably among children, complicating clinical care and return to learn and play. Persistent PCS including physical, emotional, and cognitive symptoms, result in increased school absenteeism, social isolation, and psychological distress. Early PCS diagnosis and access to evidence-based return-to-health and -school interventions are strongly linked to positive health and academic outcomes. Yet models to identify children at high risk for persistent PCS are lacking. PCS have been linked to inflammatory processes occurring within the injured brain. Preliminary evidence suggests that fatigue, another symptom likely contributing to poor outcomes, is also a biological byproduct of pediatric concussions. Importantly, even though 73% of children report continuous fatigue after concussion, this symptom is rarely studied along with other PCS. Prior research has focused on the relationship between inflammatory biomarkers and PCS severity but has not examined this relationship longitudinally. Acute symptom severity alone, however, is a poor prognostic of clinical outcomes in concussed children. Symptom severity immediately postinjury does not explain why at least 25% of children still experience PCS after 1 year or why even children who may appear asymptomatic still report academic and social challenges months after concussion. To identify which children are at high risk for persistent PCS and poor health, academic, and social outcomes, research tracking PCS trajectories and describing school-based impacts across the entire first year postinjury is critically needed. This proposal will 1) define novel PCS trajectory typologies in a racially/ethnically diverse population of 500 children with concussion (11-17 years, near equal distribution by sex), 2) identify associations between these typologies and patterns of inflammatory biomarkers, 3) develop a risk stratification model to identify children at risk for persistent PCS; and 4) gain unique insights and describe PCS impact, including fatigue, on longer-term academic and social outcomes. We will be the first to use NIH's symptom science model and patient-reported outcomes to explore the patterns of fatigue and other physical, cognitive, psychological, emotional and academic responses to concussion in children over a full year. Our model will enable clinicians and educators to identify children most at risk for poor long-term health, social, and academic outcomes after concussion. This work is critical to meeting our long-term goal of developing personalized concussion symptom management strategies to improve outcomes and reduce disparities in the health and quality of life of children.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with concussion that occurred within the past 7 days
* Glasgow Coma Scale (GCS) score between 13-15
* English speaking

Exclusion Criteria:

* Diagnosed with moderate or severe traumatic brain injury
* Polytrauma
* Nontraumatic brain injury
* Pregnancy

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Subjects will be recruited from concussion clinics in the Raleigh-Durham metro area of North Carolina.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-05-23 (Actual); Primary Completion 2028-02-28 (Estimated); Study Completion 2028-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in concussion symptom burden and severity as measured by the Post Concussion Symptom Scale (PCSS) | Within 7 days of injury, 30 days post injury, 90 days post injury, 180 days post injury, 270 days post injury and 360 days post injury
  The PCSS consists of 22 questions that relate to post-concussive symptoms. Survey-takers are asked to rate each symptom according to a 7-point Likert scale ranging from 0-6. Higher scores indicate a higher severity of post-concussive symptoms. The greatest possible score is 132 and the lowest possible score is 0.
Change in post concussion fatigue burden and severity as measured by the PROMIS Pediatric Item Bank v2.0 - Fatigue | Within 7 days of injury, 30 days post injury, 90 days post injury, 180 days post injury, 270 days post injury and 360 days post injury
  The PROMIS Pediatric Fatigue item bank consists of 25 self-report items which measure fatigue symptoms in children aged 8-17 years. Items are ranked on a 5-point likert scale ranging from 1 (Never) to 5 (Almost Always). Raw scores are converted to T-scores using scoring tables. A T-score of 50 is the average for the United States general population. A higher PROMIS T-score represents more of the concept being measured. For negatively-worded concepts like fatigue, a T-score of 60 is one SD worse greater degree of fatigue than average. By comparison, a fatigue T-score of 40 is one SD better lesser degree of fatigue than average.
Change in degree of involvement with one's peers in usual social roles, activities and responsibilities as measured by the Neuro-QoL Item Bank v1.0 - Pediatric Social Relations - Interaction with Peers | Within 7 days of injury, 30 days post injury, 90 days post injury, 180 days post injury, 270 days post injury and 360 days post injury
  This instrument consists of 8 self-report items focused on patient-reported involvement with peers in usual social roles, activities, and responsibilities. Items are rated on a 5-point likert scale ranging from 1 (Never Interacting) to 5 (Always Interacting). Raw scores are converted to T-scores using conversion tables, with a T-score of 50 as the mean. A higher Neuro-QoL T-score represents more of the concept being measured. For positively-worded concepts this measure, a T-score of 40 is one SD worse less interaction with peers than average. By comparison, a fatigue T-score of 60 is one SD better more interaction with peers than average.
Change in perceived difficulties in everyday cognitive abilities such as memory, attention, concentration, processing speed and organization skill as measured by the Neuro-QoL Item Bank v2.0 - Pediatric Cognitive Function | Within 7 days of injury, 30 days post injury, 90 days post injury, 180 days post injury, 270 days post injury and 360 days post injury
  This instrument consists of 8 self-report items focused on patient-reported difficulties with basic cognitive abilities such as memory, attention, concentration, processing speed, and organization skill. Items are rated on a 5-point likert scale ranging from 1 (Not at all) to 5 (Very much). Raw scores are converted to T-scores using conversion tables, with a T-score of 50 as the mean. A higher Neuro-QoL T-score represents more of the concept being measured. For cognitive function, a T-score of 40 is one SD less difficulty than average. By comparison, a T-score of 60 is one SD more difficulty than average .
Change in academic needs of a student following concussion as measured by the Concussion Learning Assessment & School Survey, 3rd Edition (CLASS-3) | Within 7 days of injury, 30 days post injury, 90 days post injury, 180 days post injury, 270 days post injury and 360 days post injury
  This measure consists of four scale scores (General Academic Concern, Academic Problems, School Stresses, and Academic Subjects) and a cumulative score is generated for each of the 4 scales [0-3 - General Academic Concern (1 item, total score range 0-3), Academic Problems (14 items, total score range 0-42), School Stresses (6 items, total score range 0-6); 0-4 - Academic Subjects (4 items, total score range 0-16)], which in sum can be considered as a clinical measure to assess and monitor the academic needs of a student following concussion. Higher scores correlate with greater difficulty with academic needs.
Salivary Interferon Gamma | Within 7 days of injury, 30 days post injury, 90 days post injury, 180 days post injury, 270 days post injury and 360 days post injury
  Salivary levels of inflammatory cytokine associated with post concussive symptoms
Salivary Interleukin-1 Beta | Within 7 days of injury, 30 days post injury, 90 days post injury, 180 days post injury, 270 days post injury and 360 days post injury
  Salivary levels of inflammatory cytokine associated with post concussive symptoms
Salivary Interleukin-6 | Within 7 days of injury, 30 days post injury, 90 days post injury, 180 days post injury, 270 days post injury and 360 days post injury
  Salivary levels of inflammatory cytokine associated with post concussive symptoms
Salivary Interleukin-8 | Within 7 days of injury, 30 days post injury, 90 days post injury, 180 days post injury, 270 days post injury and 360 days post injury
  Salivary levels of inflammatory cytokine associated with post concussive symptoms
Salivary Interleukin-10 | Within 7 days of injury, 30 days post injury, 90 days post injury, 180 days post injury, 270 days post injury and 360 days post injury
  Salivary levels of inflammatory cytokine associated with post concussive symptoms
Salivary TNF-Alpha | Within 7 days of injury, 30 days post injury, 90 days post injury, 180 days post injury, 270 days post injury and 360 days post injury
  Salivary levels of inflammatory cytokine associated with post concussive symptoms
Pubertal status | Within 7 days of injury, 30 days post injury, 90 days post injury, 180 days post injury, 270 days post injury and 360 days post injury
  Salivary DHEA concentration
  The high levels of DHEA that are secreted beginning in mid-childhood (~8 years of age) serve as a marker of adrenarche (puberty). DHEA level rises before external physical changes of puberty become obvious. Levels of DHEA in saliva have been shown to be a reliable index of blood levels in children and adolescents and are not dependent on time of day. DHEA age/sex-based reference ranges will be used to determine pubertal maturation. The assay results range from 10.2 pg/mL to 1000 pg/mL with higher levels correlating with later Tanner stages of puberty.
Presence of genetic variants in genes that code for inflammatory cytokines | Within 7 days of injury
  Inflammatory genetic variants involved in brain injury and in fatigue in the following genes:
  APOE, IGSF3, IFN-γ, IL-1β, IL-6, IL-8, IL-10, MAPT, TNF-α, TNFAIP1, TNFAIP8

CONTACTS AND LOCATIONS:
Overall Officials: Karin Reuter-Rice, PhD, Principal Investigator — Duke University School of Nursing
Locations (1):
- Duke University Health System, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reuter-Rice K, Fitterer AN, Duquette P, Yang Q, Palipana AK, Laskowitz D, Garrett ME, Fletcher M, Smith J, Makor L, Grant G, Ramsey K, Bloom OJ, Ashley-Koch AE. A study protocol for risk stratification in children with concussion (RSiCC): Theoretical framework, design, and methods. PLoS One. 2024 Jul 18;19(7):e0306399. doi: 10.1371/journal.pone.0306399. eCollection 2024. PMID 39024215